CLINICAL TRIAL: NCT03459859
Title: An Open-Label, Dose Escalation, Phase 1 Study of PEVONEDISTAT, a Novel Inhibitor of the NEDD8-Activating Enzyme (NAE), in Combination With Low Dose Cytarabine (LDAC) in Adult Patients With Acute Myelogenous Leukemia (AML) and Advanced Myelodysplastic Syndromes (MDS)
Brief Title: Pevonedistat and Low Dose Cytarabine in Adult Patients With AML and MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Justin Watts, MD (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Justin Watts, MD, Assistant Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180054; NCI-2019-06910 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2018-03-03; First posted 2018-03-09 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Acute Myelogenous Leukemia; AML; Advanced Myelodysplastic Syndromes; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pevonedistat; Cytarabine

STUDY DESIGN:
Intervention Model Description: Dose escalation, traditional 3:3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pevonedistat 10 LDAC 20 (Experimental): Dose Level -1: Pevonedistat 10 mg/m2, low dose Cytarabine (LDAC) 20 mg/m2 for up to 16 cycles of 28 days each, per protocol
  Interventions: Drug: Pevonedistat; Drug: Cytarabine
- Pevonedistat 15 LDAC 20 (Experimental): Dose Level 1 (Starting Dose): Pevonedistat 15 mg/m2, low dose Cytarabine (LDAC) 20 mg/m2 for up to 16 cycles of 28 days each, per protocol
  Interventions: Drug: Pevonedistat; Drug: Cytarabine
- Pevonedistat 20 LDAC 20 (Experimental): Dose Level 2: Pevonedistat 20 mg/m2, low dose Cytarabine 20 mg/m2 for up to 16 cycles of 28 days each, per protocol
  Interventions: Drug: Pevonedistat; Drug: Cytarabine
- Pevonedistat 25 LDAC 20 (Experimental): Dose Level 3: Pevonedistat 25 mg/m2, low dose Cytarabine (LDAC) 20 mg/m2 for up to 16 cycles of 28 days each, per protocol
  Interventions: Drug: Pevonedistat; Drug: Cytarabine

INTERVENTIONS:
Drug: Pevonedistat — Administered intravenous (IV) infusion over one hour on Days 1, 3 and 5 of each cycle, after administration of LDAC per protocol.
  Other Names: MLN4924
Drug: Cytarabine — Low dose Cytarabine (LDAC) administered subcutaneously (SC) daily for 10 days of every 28-day cycle.
  Other Names: ara-C

SUMMARY:
The investigators hypothesize that the combination of Pevonedistat/Low-Dose Cytarabine (LDAC) therapy will be tolerable, that a recommended phase 2 dose of Pevonedistat in combination with LDAC will be identified, and that the combination therapy will show evidence of clinical activity in adult patients with Relapsed/Refractory Acute Myelogenous Leukemia (AML) and Advanced Myelodysplastic Syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

A. Confirmed diagnosis of one of the following:

1. Relapsed/refractory Acute Myelogenous Leukemia (AML) where no alternative life prolonging therapy exists. Treatment naïve patients may also be considered eligible if in the opinion of the investigator, these patients are unlikely to benefit from alternative therapy (eg conventional chemotherapy, hypomethylating agents).
2. Relapsed/refractory Myelodysplasic Syndrome (MDS) following at least two courses of a hypomethylating agent (eg azacitidine or decitabine). Patients intolerant of hypomethylating agents (irrespective of the number of cycles administered) will also be considered eligible. MDS eligibility limited to patients with intermediate, high or very high risk based on IPSS-R.

B. Adult male or female patients 18 years of age or older.

C. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2

D. Patients must satisfy the following laboratory criteria:

1. Albumin > 2.7 g/dL
2. Total bilirubin ≤ upper limit of normal (ULN) except in patients with Gilbert's syndrome. Patients with Gilbert's syndrome may enroll if direct bilirubin ≤1.5 x ULN of the direct bilirubin
3. Alanine transaminase (ALT) and Aspartate transaminase (AST) must be ≤ 2.5 × ULN
4. Creatinine 1.5 x ULN or calculated creatinine clearance > 50ml/min
5. Hemoglobin > 8 g/dL (prior red blood cell (RBC) transfusion allowed). Patients may be transfused to achieve this value. Elevated indirect bilirubin due to post-transfusion hemolysis is allowed.
6. White blood cell (WBC) count < 50,000/µL before administration of PEVONEDISTAT on Cycle 1 Day 1. Note: Hydroxyurea may be used to control the level of circulating leukemic blast cell counts to not lower than 10,000/µL during the study.

E. Suitable venous access to allow for all study related blood sampling (safety and research).

F. Estimated life expectancy, in the judgment of the Investigator, which will permit receipt of at least 6 weeks of treatment.

G. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

H. Female patients who:

1. Are postmenopausal (see Appendix for definition) for at least 1 year before the screening visit, OR
2. Are surgically sterile, OR
3. If they are of childbearing potential:

   * Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception).

I. Male patients, even if surgically sterilized (ie, status postvasectomy), who:

1. Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception).

J. Able to undergo bone marrow aspiration at screening.

Exclusion Criteria:

A. Treatment with clinically significant metabolic enzyme inducers within 14 days before the first dose of the study drug. Strong CYP3A inhibitors and CYP3A inducers are not permitted during the study.

B. Therapy with any investigational products, anti-neoplastic therapy, or radiotherapy within 14 days prior to Cycle 1 Day 1. Patients actively receiving hydroxyurea are eligible and may continue to receive hydroxyurea during protocol treatment.

C. Candidates for standard and/or potentially curative treatments (a candidate is defined as a patient that is both eligible and willing to have these treatments)

D. Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period.

E. Grade 2 or higher diarrhea as defined by NCI CTCAE Version 4.03 despite optimal anti-diarrheal supportive care within 7 days prior to Cycle1 Day1.

F. Known cardiopulmonary disease defined as one of the following:

1. Uncontrolled high blood pressure (ie, systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg).
2. Cardiomyopathy or history of ischemic heart disease; patients with ischemic heart disease who have had acute coronary syndrome (ACS), MI, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll;
3. Clinically significant arrhythmia including:,history of polymorphic ventricular fibrillation or torsade de pointes); permanent atrial fibrillation [a fib], defined as a fib for ≥6 months; persistent a fib, defined as sustained afib >7 days and/or requiring cardioversion in the 4 weeks before screening; Grade 3 a fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation. Patients with paroxysmal a fib are permitted to enroll. However, patients with < Grade 3 atrial fibrillation (a fib) for a period of at least 6 months may enroll provided that their rate is controlled on a stable regimen.
4. Implantable cardioverter defibrillator;
5. Congestive heart failure (New York Heart Association (NYHA) Class III or IV; or Class II with a recent decompensation requiring hospitalization or referral to a heart failure clinic within 4 weeks before screening), myocardial infarction and/or revascularization (eg, coronary artery bypass graft, stent) within 6 months of first dose of study drug.
6. Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing);
7. Pulmonary hypertension.
8. Patients with Grade 2 or higher prolonged rate corrected QT (QTc) interval (≥ 481msec), calculated according to institutional guidelines.
9. Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography - LVEF assessment is not required for screening, and will only be done at the investigators discretion if clinically indicated..
10. Known moderate to severe chronic obstructive pulmonary disease (COPD), interstitial lung disease, and pulmonary fibrosis.

G. Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia.

H. Known human immunodeficiency virus (HIV) seropositive.

I. Known hepatitis B surface antigen seropositive (Note: Patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.)

J. Known or suspected active hepatitis C infections (Patients who are hepatitis C surface antigen-positive are eligible).

K. Females of child bearing potential who refuse to either practice 2 effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 30 days after the last dose of study drug.

L. Males of child bearing potential who refuse to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug. (Includes males surgically sterilized - i.e. status post vasectomy).

M. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.

N. Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).

O. Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).

P. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.

Q. Symptomatic central nervous system (CNS) involvement.

R. Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.

S. Known hepatic cirrhosis or severe pre-existing hepatic impairment.

T. Systemic anti-neoplastic therapy or radiotherapy within 14 days before the first dose of any study drug, except for hydroxyurea.

U. Patients with uncontrolled coagulopathy or bleeding disorder.

V. Life-threatening illness unrelated to cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Safety Profile of Combination Pevonedistat/LDAC Therapy: Rate of Toxicity in Study Participants | From Cycle 1 Day 1 to End of Study, up to 18 months
  Rate of toxicity in study participants receiving at least one dose of combination Pevonedistat/LDAC protocol therapy, including determination of dose limiting toxicities (DLTs), serious adverse events (SAEs), and AEs. Toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03.
Maximum Tolerated Dose (MTD) and Recommended Phase 2 (RP2D) Dose of Pevonedistat in Combination with Low Dose Cytarabine (LDAC) | From Cycle 1 Day 1 to End of Study, up to 18 months
  Determination of the MTD and RP2D of PEVONEDISTAT administered intravenously in patients with AML and advanced MDS when given in combination with low dose cytarabine (LDAC).

SECONDARY OUTCOMES:
Rate of Efficacy in Study Participants | Up to 17 months
  Rate of complete response (CR) and partial response (PR) in study participants to Pevonedistat/LDAC combination therapy. Response will be determined using serial blood and bone marrow sampling throughout the course of treatment, and assessed according to revised/modified International Working Group (IWG) Response Criteria - Cheson et al. 2003 for AML and Cheson et al. 2006 for MDS.
  Morphologic complete remission (CR), cytogenetic CR, and molecular CR will be assessed based on blood counts, marrow blast percentage, cytogenetic studies and mutational analysis on every occasion the bone marrow is examined to assess for response.
Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of Pevonedistat | Cycle 1 Days 1, 2 3, and 5
  Pharmacokinetic effects of IV-administered PEVONEDISTAT in plasma will be measured when combined with LDAC. Cmax is the maximum (or peak) plasma concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose. Pharmacokinetics (PK) parameters will be determined using serial blood sampling at specified time points to determine PK effects of PEVONEDISTAT in plasma when combined with LDAC. Non-compartmental methods of analysis will be used to determine PEVONEDISTAT PK parameters following IV dosing of patients in Cycle 1.
Pharmacokinetics (PK): Time to Cmax (Tmax) of Pevonedistat | Cycle 1 Days 1, 2, 3, and 5
  Pharmacokinetic effects of IV-administered PEVONEDISTAT in plasma will be measured when combined with LDAC. Tmax is the time it takes a drug or other substance to reach the maximum concentration (Cmax). Pharmacokinetics (PK) parameters will be determined using serial blood sampling at specified time points to determine PK effects of PEVONEDISTAT in plasma when combined with LDAC. Non-compartmental methods of analysis will be used to determine PEVONEDISTAT PK parameters following IV dosing of patients in Cycle 1.
Pharmacokinetics (PK): Area Under the Plasma Concentration-Time curve from time 0 to 24 hours post-dose of Pevonedistat (AUC24hr). | Cycle 1 Days 1, 2, 3, and 5
  Pharmacokinetic effects of IV-administered PEVONEDISTAT in plasma will be measured when combined with LDAC. The area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC24hr) will be assessed. Pharmacokinetics (PK) parameters will be determined using serial blood sampling at specified time points to determine PK effects of PEVONEDISTAT in plasma when combined with LDAC. Non-compartmental methods of analysis will be used to determine PEVONEDISTAT PK parameters following IV dosing of patients in Cycle 1.
Pharmacokinetics (PK): Terminal disposition phase half-life (t1/2) of Plasma Concentration of Pevonedistat | Cycle 1 Days 1, 2, 3, and 5
  Pharmacokinetic effects of IV-administered PEVONEDISTAT in plasma will be measured when combined with LDAC. Terminal phase half-life (t1/2) will be assessed. Half-life (t1/2) is the amount of time it takes for the drug concentration in the plasma to decline by half. Pharmacokinetics (PK) parameters will be determined using serial blood sampling at specified time points to determine PK effects of PEVONEDISTAT in plasma when combined with LDAC. Non-compartmental methods of analysis will be used to determine PEVONEDISTAT PK parameters following IV dosing of patients in Cycle 1.
Pharmacodynamics (PD): Induction Levels of CRL substrates | Baseline, Cycle 1 Days 1, 2, and 5; and End of Study, up to 18 months (+/- 10 days)
  Pharmacodynamics (PD) measurements will be obtained from serial blood and bone marrow sampling at specified time points to describe the PD effects of PEVONEDISTAT when combined with LDAC. The following endpoints will be analyzed: Induction of Cullin Ring Ligase (CRL) substrates by immunoblotting (e.g. nuclear factor (erythroid-derived 2)-like 2 (NRF2), chromatin licensing and DNA replication factor 1 (CDT1), pIKB and others).
Pharmacodynamics (PD): Induction Levels of Pathway Markers | Baseline, Cycle 1 Days 1, 2, and 5; and End of Study, up to 18 months (+/- 10 days)
  Pharmacodynamics (PD) measurements will be obtained from serial blood and bone marrow sampling at specified time points to describe the PD effects of PEVONEDISTAT when combined with LDAC. The following endpoints will be analyzed: Induction of pathway markers (eg SQ01 by polymerase chain reaction (PCR) in peripheral blood mononuclear cells) as well as other known indicators of pathway inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Watts, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No